CLINICAL TRIAL: NCT01609634
Title: A Randomised, Controlled, Double-blind Trial to Investigate the Effects of a New Infant Formula in Healthy Term Subjects on Growth, Body Composition, Tolerance and Safety.
Brief Title: New Infant Formula Trial in Healthy Term Subjects on Growth, Body Composition, Tolerance and Safety
Acronym: Venus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EBB15GL04184
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Healthy; Term infants; Growth; Body composition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Key Group of interest (Active Comparator): Subjects who started test product / control product 1 / control product 2 by 1-month of age
  Interventions: Other: Test Product
- Other-fed Group (Active Comparator): Subjects who started test product / control product 1 / control product 2 and continued on breast-feeding
  Interventions: Other: Control Product 1
- Breast Fed Reference Group (Active Comparator): Subjects who are exclusively breast-fed up to 4 months of age and not started on test product / control product 1 / control product 2.
  Interventions: Other: Control Product 2

INTERVENTIONS:
Other: Test Product — Standard infant formula/follow-on formula with added scGOS/lcFOS and Nuturis®
  Arms: Key Group of interest
Other: Control Product 1 — Control group 1: Standard infant formula/follow-on formula with added scGOS/lcFOS
  Arms: Other-fed Group
Other: Control Product 2 — Control group: Standard infant formula/follow-on formula with standard fat droplets and without specific prebiotic oligosaccharides.
  Arms: Breast Fed Reference Group

SUMMARY:
This study is initiated to investigate the effect of a new infant formula in healthy term subjects on growth, body composition, tolerance and safety.

DETAILED DESCRIPTION:
This is a "best after breast design" to measure the effect of this new infant formula in healthy term subjects on growth, body composition, tolerance and safety including immune status, gut microbiota, and early indicators (markers) of disease. These markers will be explored if they could predict the risk of eczema and other allergic disease, and to evaluate if these markers are influenced by early nutrition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infants (gestational age ≥ 37 and ≤ 42 weeks)
2. Age ≤ 28 days
3. Birth weight within normal range for gestational age and sex (3rd to 90th percentile according to applicable growth charts)
4. Head circumference at birth within normal range (3rd to 90th percentile of the chart)
5. Chinese, Malay, or Indian ethnicity
6. Written informed consent from parent(s)
7. Currently reside in Singapore and with the intention to reside in Singapore for at least the next 2 years

Exclusion criteria for the pregnant women/parents:

1. Pregnant women / mothers who are currently participating or will participate in any other (clinical) study involving investigational or marketed products during pregnancy and/or lactation.
2. Pregnant women / mothers known to suffer from hepatitis B or human immunodeficiency virus (HIV)
3. Pregnant women / mothers known to have other significant medical condition (including during pregnancy) that might interfere with the study or known to affect intra-uterine growth (including, but not limited to: placenta previa, pre-eclampsia, eclampsia, gestational diabetes requiring insulin or oral medication), as per investigator's clinical judgement
4. Incapability of the parents to comply with study protocol or Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements

   Exclusion criteria for the subjects:
5. Infants known to have current or previous illnesses/ conditions or intervention which could interfere with the study (growth), as per investigator's clinical judgement
6. Infants with known congenital diseases or malformations which could interfere with the study (e.g. gastrointestinal malformations, congenital immunodeficiency), as per investigator's clinical judgement
7. Infants who need to be fed with a special diet other than a standard cow's milk-based infant formula
8. Infants who received any other infant formula, except the infant formula given in between birth and the initial breast-feeding (maximum of 3 consecutive days)
9. Infants with any history of or current participation in any other study involving investigational or marketed products.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 541 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Weight gain per day | 17 weeks
  Weight gain per day from randomisation until 17 weeks of age.
Total weight gain | 12 months
  Total weight gain from birth until 12 months of age
Sum of skin fold thicknesses | 24 months
  Sum of skin fold thicknesses: triceps, biceps, suprailiac, subscapular until 24 months of age in subjects receiving the test product 1, test product 2, or control product.

SECONDARY OUTCOMES:
Recumbent length, head circumference, mid-upper arm circumference, skin folds | 17 weeks
  Recumbent length, head circumference, mid-upper arm circumference, skin folds gain per day for subjects receiving test product 1 or test product 2
Skin-fold thickness | 12 months
  Sum of four Skin-fold thickness: triceps, biceps, subscapular and suprailiac measured until 12 months of age
Weight, length, BMI, head circumference, mid-upper arm circumference, subscapular skinfold, triceps skinfold | 24 months
  Weight, length, BMI, head circumference, mid-upper arm circumference, subscapular skinfold, triceps skinfold measured until 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Oon Hoe Teoh, Dr, MD, Principal Investigator — KK Women's and Children's Hospital; Yap Seng Chong, A/Prof, MD, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Merwe LF, Mulder KA, van Oudenhoven FM, Shek LP, Teoh OH, Pang WW. Mixed Milk Feeding Patterns and Growth Outcomes During the First Year of Life in Asian Infants: Application of Predefined Feeding Clusters to Test Associations. Curr Dev Nutr. 2025 Oct 3;9(11):107565. doi: 10.1016/j.cdnut.2025.107565. eCollection 2025 Nov. PMID 41189742